CLINICAL TRIAL: NCT01229306
Title: Repeat Ablation Procedure in Patients With Relapse of Paroxysmal Atrial Fibrillation Using Reisolation of Pulmonary Vein Versus Reisolation of Pulmonary Vein With Additional Anterior Line
Brief Title: Repeat Ablation Procedure in Patients With Relapse of Atrial Fibrillation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Deutsches Herzzentrum München, Abteilung Elektrophysiologie
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GER-EP-002
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-05

CONDITIONS: Ablation; Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- reisolation of all PV and additional anterior line (Experimental)
  Interventions: Procedure: Ablation
- reisolation of all pulmonary veins (Placebo Comparator)
  Interventions: Procedure: Ablation

INTERVENTIONS:
Procedure: Ablation — Ablation of atrial fibrillation

SUMMARY:
Catheter ablation with isolation of the pulmonary veins has proven to be an effective treatment option in patients with paroxysmal atrial fibrillation. In patients who have a relapse of paroxysmal atrial fibrillation after one ablation procedure the investigators compare the reisolation of all pulmonary veins to reisolation plus an anterior left atrial line.

DETAILED DESCRIPTION:
Catheter ablation with isolation of the pulmonary veins has proven to be an effective treatment option in patients with paroxysmal atrial fibrillation. In patients who have a relapse of paroxysmal atrial fibrillation after one ablation procedure we compare the reisolation of all pulmonary veins to reisolation plus an anterior left atrial line.

ELIGIBILITY:
Inclusion Criteria:

* relapse of atrial fibrillation

Exclusion Criteria:

* contraindication for ablation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-07 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Freedom of atrial arrhythmias

SECONDARY OUTCOMES:
Quality of life, number of reconnected pulmonary veins, safety

CONTACTS AND LOCATIONS:
Locations (1):
- Deutsches Herzzentrum, München, Bayer, Germany